CLINICAL TRIAL: NCT04580940
Title: Flexible Percutaneous Transhepatic Cholangiopancreatoscopy (PTCS) in Complex Pancreaticobiliary Disease
Brief Title: SpyGlass™ Discover Percutaneous
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: E7160
Record Dates: First submitted 2020-09-23; First posted 2020-10-09 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Pancreatic Diseases; Bile Duct Obstruction; Bile Duct Diseases
Keywords: Percutaneous transhepatic cholangiopancreatoscopy; spyglass discover; pancreaticobiliary disease
MeSH Terms: conditions — Pancreatic Diseases; Cholestasis; Bile Duct Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Subjects with complex pancreaticobiliary disease: All subjects will undergo the percutaneous transhepatic cholangiopancreatoscopy with the SpyGlass Discover System.
  Interventions: Device: SpyGlass™ Discover Digital System

INTERVENTIONS:
Device: SpyGlass™ Discover Digital System — Observational, prospective, registry study for the clinical utility of the SpyGlass Discover digital catheter during a PTCS procedure.

SUMMARY:
To document the clinical utility of percutaneous cholangiopancreatoscopy using a thin, disposable, flexible endoscope for evaluation and treatment of complex pancreaticobiliary disease in a prospective, multi-center case series

DETAILED DESCRIPTION:
This case series aims to illustrate the clinical utility of percutaneous transhepatic cholangiopancreatoscopy using a thin, disposable, flexible endoscope performed by gastroenterological endoscopists and/or interventional radiologists in procedures including but not limited to:

* PTCS for tissue diagnosis in cases of surgically or pathologically-altered anatomy,
* PTCS for stone removal after surgically or pathologically-altered anatomy,
* Percutaneous rendezvous to aid ERCP after failed endoscopic cannulation,
* Percutaneous delivery of palliative intraluminal brachytherapy,
* Intra-procedural percutaneous salvage procedures when an initial route of access fails

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled for a percutaneous transhepatic procedure to access the pancreaticobiliary anatomy that will accommodate passage of SpyGlass™ Discover Digital Catheter per local standard of practice
2. Written informed consent from patient or legally authorized representative of the patient

Exclusion Criteria:

1. Contraindication for cholangiopancreatoscopy
2. Subjects with unresolved adverse event(s) associated with prior percutaneous pancreaticobiliary ductal access
3. <18 years of age
4. Potentially vulnerable subjects, including, but not limited to pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with complex pancreaticobiliary disease
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-07-27 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2023-01-14 (Actual)

PRIMARY OUTCOMES:
Achieving clinical intent of procedure as indicated | 1 month
  Physicians will report achieving clinical success by recording the completed procedures compared to procedures planned by 30 days (+/- 3 days) after index PTCS.

SECONDARY OUTCOMES:
Number of Adverse Events | 1 month
  Serious adverse events related to the study device, accessory devices used through the working channel of the SpyGlass™ Discover Digital Catheter or the cholangiopancreatoscopy portion of the PTCS procedure(s).
Technical success | During index procedure
  Rate at which SpyGlass™ Discover digital catheter can be advanced to the target lesion or stone(s) and visualize the target
Procedural Time | During index procedure
  Time elapsed between first insertion to last removal of the SpyGlass™ Discover digital catheter
Number of PTCS procedures | 1 month
  Number of PTCS procedures required to achieve clinical success until the end of follow-up
Endoscopist rating | During index procedure
  Endoscopist rating of the following attributes when using SpyGlass™ Discover Digital Catheter compared to marketed reusable scopes Ability to complete the procedure Ability to retroflex Ability to selectively advance into targeted ducts Ability to obtain targeted biopsies Ability to grasp stones Ability to guide lithotripsy Ability to suction Ability to irrigate Ability to advance accessories through scope channel Image quality

CONTACTS AND LOCATIONS:
Overall Officials: Ivo Boskoski, MD, PhD, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS; Torsten Beyna, MD, PhD, Principal Investigator — Evangelisches Krakenhaus Düsseldorf; Mehran Fotoohi, MD, PhD, Principal Investigator — Virginia Mason; Arnaud Lemmers, MD, PhD, Principal Investigator — Erasme University Hospital; James Lau, MD, PhD, Principal Investigator — Prince of Wales Hospital; Eran Shlomovitz, MD, PhD, Principal Investigator — Toronto General Hospital, University Health Network; Mohan Ramchandani, MD, PhD, Principal Investigator — Asian Institute of Gastroenterology
Locations (7):
- Virginia Mason Medical Center, Seattle, Washington, United States
- Erasme University Hospital, Brussels, Belgium
- Toronto General Hospital, University Health Network, Toronto, Ontario, Canada
- Evangelisches Krakenhaus Düsseldorf, Düsseldorf, Germany
- Prince of Wales Hospital, Shatin, NewTerritories, Hong Kong
- Asian Institute of Gastroenterology, Hyderabad, Somajiguda, India
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, Italy

REFERENCES:
- [Derived] Boskoski I, Beyna T, Lau JY, Lemmers A, Fotoohi M, Ramchandani M, Pontecorvi V, Peetermans J, Shlomovitz E. Efficacy and safety of a single-use cholangioscope for percutaneous transhepatic cholangioscopy. Endosc Int Open. 2024 Aug 23;12(8):E981-E988. doi: 10.1055/a-2366-2265. eCollection 2024 Aug. PMID 39184059
- [Derived] Aihara H, Othman MO, Jawaid SA, Gorgun E, Sharma NR, Siddiqui UD, Peetermans JA, Rousseau MJ, Nishimura M. A multicenter, retrospective study of a through-the-needle injection-capable electrosurgical knife for endoscopic submucosal dissection. Gastrointest Endosc. 2024 Dec;100(6):1034-1042. doi: 10.1016/j.gie.2024.06.011. Epub 2024 Jun 13. PMID 38879045